CLINICAL TRIAL: NCT06435104
Title: Effects of Aromatherapy on Anxiety and Tumor Immunity of Early Breast Cancer Patients,a Pilot Study
Brief Title: Aromatherapy in the Treatment of Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-063-02
Record Dates: First submitted 2024-03-13; First posted 2024-05-30 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Early Breast Cancer
Keywords: Early breast Cancer; Anxiety; Aromatherapy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders | interventions — Neoadjuvant Therapy; Aromatherapy

STUDY DESIGN:
Intervention Model Description: The research model consists of two arms#
  1. armA:neoadjuvant chemotherapy
  2. armB:neoadjuvant chemotherapy+aromatherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant chemotherapy (Other): Patients will receive effective neoadjuvant chemotherapy for at least 2 courses.
  Interventions: Other: neoadjuvant chemotherapy
- neoadjuvant chemotherapy+aromatherapy (Experimental): Patients will receive effective neoadjuvant chemotherapy for at least 2 courses, and the aromatherapy is recommended to continue throughout neoadjuvant chemotherapy.
  Interventions: Other: neoadjuvant chemotherapy; Other: aromatherapy

INTERVENTIONS:
Other: neoadjuvant chemotherapy — The neoadjuvant chemotherapy plan will be selected according to the recommendations of the NCCN guidelines and the Chinese CSCO guidelines for early breast cancer.The neoadjuvant chemotherapy plans include:AC-T(HP),TCb(HP),AC-TCb, in which A represents anthracycline, C represents cyclophosphamide, T represents taxane, Cb represents carboplatin, H represents trastuzumab, and P represents pertuzumab.
Other: aromatherapy — Patients will inhale essential oils during the neoadjuvant chemotherapy courses.
  Arms: neoadjuvant chemotherapy+aromatherapy

SUMMARY:
Breast cancer is a major threat to women's health, and chemotherapy is one of the most important treatment method. Chemotherapy is cytotoxic , and has a positive tumor immune effect. However, it is worth noting that anxiety caused by breast cancer itself and adverse reactions of chemotherapy not only affects the patients' quality of life, but also reduces the treatment compliance and even survival benefits of patients. Previous literatures have shown that aromatherapy may improve chemotherapy-induced anxiety and even affect anti-tumor immunity.

Therefore,we envisage that aromatherapy conbimed with chemotherapy in the treatment of breast cancer in clinical practice has the advantages of improving efficacy and survival.

However, there is still a lack of relevant clinical studies. We planned to design a prospective clinical trial to evaluate the efficacy and safety of aromatherapy combined with chemotherapy on anxiety, relevant sympathetic neurotransmitters and tumor immunity in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women all over the world. In China, the incidence of breast cancer is increasing, especially in the economically developed cities. Studies have shown that the breast cancer patients have a higher incidence of anxiety and depression to the general population. Tumor burden is an important chronic stressor that can cause a wide range of negative emotions, such as anxiety and depression. According to the data published by the World Health Organization, the incidence of depression in cancer patients is between 20% to 45%, which is far more than the incidence of 6.1% to 9.5% in the general population.Among them, the depression tendency of breast cancer patients is particularly obvious, and up to 80% of breast cancer patients suffer from different degrees of depression. Depression and anxiety have a crucial influence on the physiological and psychological function, treatment compliance and the quality of life of breast cancer patients, and may even be an important factor affecting the mortality of breast cancer patients.

Therefore, how to improve the anxiety of breast cancer patients to improve the quality of life and even the survival time of patients has vital clinical value. Considering the adverse reactions and tolerance of current anti-anxiety drugs, more mild and effective anti-anxiety methods are expected in clinical practice. Among them, as an important means of rehabilitation treatment, aromatherapy has obtained surprising data in the prevention of adverse reactions of chemotherapy and the improvement of insomnia, so the value of aromatherapy in the improvement of anxiety is also expected.

In conclusion, Breast cancer is a major threat to women's health, and chemotherapy is one of the most important treatment method. Chemotherapy is cytotoxic , and has a positive tumor immune effect. However, it is worth noting that anxiety and depression caused by breast cancer disease itself and adverse reactions of chemotherapy not only affects the quality of life of patients, but also reduces the treatment compliance and even survival benefits of patients. Previous literatures have shown that aromatherapy may improve chemotherapy-induced anxiety and even have influence on tumor immunity. However, there is still lack of relevant clinical researches. Therefore, we plan to design a prospective clinical study to evaluate the effect of aromatherapy combined with neoadjuvant chemotherapy on anxiety, sympathetic neurotransmitters and tumor immunity in early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (age 18-80 years) with early breast cancer confirmed by pathology.
2. Patients have not received any anti-tumor treatment,and are planning to receive neoadjuvant chemotherapy.
3. Patients with mild anxiety scored 50 in Self-Rating Anxiety Scale.
4. ECOG physical status score ≤ 2 and expected survival of not less than 3 months.
5. At least one measurable lesion should be present in the imaging examination within 2 weeks prior to enrollment.
6. Adequate reserve of bone marrow function: white blood cell count ≥ 3.0×10^9/L, neutrophil count ≥ 1.5 × 10^9/L; Platelet count ≥ 70 × 10^9/L.
7. Basically normal liver, kidney and cardiac function:total bilirubin≤3 times the upper limit of normal value,Alanine Transaminase/Aspartate Aminotransferase≤2.5 times the upper limit of normal value(patients with liver metastases≤5 times the upper limit of normal value)，serum creatinine≤1.5 times the upper limit of normal value or creatinine clearance rate≥60mL/min, left ventricular ejection fraction (LVEF) ≥ 55%,QTcF(Fridericia correction) ≤ 470 ms.
8. Be able to understand the research process, volunteer to participate in the study, and sign informed consent.

Exclusion Criteria:

1. Patients who are not able to receive aromatherapy:be allergic to aromatherapy materials or suffer from heterosmia.
2. Received surgery within 2 weeks prior to enrollment.
3. Patients with severe cardiovascular and cerebrovascular events within 12 months, including but not limited to unstable angina, myocardial infarction, cerebral hemorrhage, and cerebral infarction (except asymptomatic lacunar infarction requiring no treatment)
4. Patients with active autoimmune diseases requiring treatment (e.g., corticosteroids or immunosuppressive drugs) within the past 2 years. Patients who need corticosteroid replacement therapy for adrenal insufficiency were excluded.
5. Patients with a definite past medical history or present medical history of neurological or mental disorders, including epilepsy or dementia.
6. The researchers believe that patients are not suitable to participate in any other circumstances of this study, which may interfere with the accompanying diseases or conditions of the study, or have any serious medical obstacles that may affect the safety of the subjects.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety score | before neoadjuvant chemotherapy and at the end of neoadjuvant chemotherapy course 2 (each course is 21 days)
  Changes of anxiety scores (Hamilton Anxiety Scale and State-trait anxiety inventory scale) before and after two neoadjuvant chemotherapy courses.

SECONDARY OUTCOMES:
Overall Survival, OS | 2 years
  The time from the start of randomization to death due to any cause
Quality of life scale score,QoL | before neoadjuvant chemotherapy and at the end of neoadjuvant chemotherapy course 2 (each course is 21 days)
  The function or quality of a patient's physical, psychological, and social adaptability is also known as quality, which is assessed according to the EROTC C30 scale.
Pathologic complete response,pCR | 2 years
  Proportion of patients with pathologic complete response after neoadjuvant chemotherapy
Disease-free survival,DFS | 2 years
  The time from diagnosis to first recurrence or death of the patient
Complete response,CR | 2 years
  All target lesions disappeared, no new lesions appeared, and tumor markers remained normal for at least 4 weeks.
Partial response,PR | 2 years
  The sum of the maximum diameters of the target lesions is reduced by≥30%,maintained for at least 4 weeks.
Stable disease,SD | 2 years
  The sum of the maximum diameters of the target lesions is within the prescribed range of partial response and progressive disease.
Progressive disease,PD | 2 years
  The sum of the maximum diameters of the target lesions increases by at least 20%, and their absolute value of diameters increases by at least 5mm, or new lesions appear.
Objective Response Rate, ORR | 2 years
  The proportion of patients with a tumor volume reduction of ≥30% and a minimum timeframe according to accepted response evaluation criteria (e.g., RECIST version 1.1 in solid tumors), including cases of complete response (CR) and partial response (PR).
Clinical Benefit Rate, CBR | 24 weeks after enrollment
  Proportion of confirmed complete response, partial response, or stable disease ≥ 24 weeks.
Anxiety rating scale | before treatment and 3 months after the last treatment
  The scores of self-rating anxiety scale (SAS) before treatment, after each treatment and 3 months after the last treatment.
Sleep rating scale | before treatment and 3 months after the last treatment
  The scores of Pittsburgh sleep quality index(PSQI) before treatment, after each treatment and 3 months after the last treatment.
Depression scale | before neoadjuvant chemotherapy and at the end of neoadjuvant chemotherapy course 2 (each course is 21 days)
  The scores of Hamilton Depression Scale(HAMD) before treatment and after 2 times of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli J Zhao, doctorate, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
As personal information of patients is involved, we decided not to share individual participant data of patients.

REFERENCES:
- [Background] Harbeck N, Penault-Llorca F, Cortes J, Gnant M, Houssami N, Poortmans P, Ruddy K, Tsang J, Cardoso F. Breast cancer. Nat Rev Dis Primers. 2019 Sep 23;5(1):66. doi: 10.1038/s41572-019-0111-2. PMID 31548545
- [Background] Xiong SY, Wen HZ, Dai LM, Lou YX, Wang ZQ, Yi YL, Yan XJ, Wu YR, Sun W, Chen PH, Yang SZ, Qi XW, Zhang Y, Wu GY. A brain-tumor neural circuit controls breast cancer progression in mice. J Clin Invest. 2023 Dec 15;133(24):e167725. doi: 10.1172/JCI167725. PMID 37847562
- [Background] Wang X, Wang N, Zhong L, Wang S, Zheng Y, Yang B, Zhang J, Lin Y, Wang Z. Prognostic value of depression and anxiety on breast cancer recurrence and mortality: a systematic review and meta-analysis of 282,203 patients. Mol Psychiatry. 2020 Dec;25(12):3186-3197. doi: 10.1038/s41380-020-00865-6. Epub 2020 Aug 20. PMID 32820237
- [Background] Carreira H, Williams R, Funston G, Stanway S, Bhaskaran K. Associations between breast cancer survivorship and adverse mental health outcomes: A matched population-based cohort study in the United Kingdom. PLoS Med. 2021 Jan 7;18(1):e1003504. doi: 10.1371/journal.pmed.1003504. eCollection 2021 Jan. PMID 33411711
- [Background] Sharma M, Grewal K, Jandrotia R, Batish DR, Singh HP, Kohli RK. Essential oils as anticancer agents: Potential role in malignancies, drug delivery mechanisms, and immune system enhancement. Biomed Pharmacother. 2022 Feb;146:112514. doi: 10.1016/j.biopha.2021.112514. Epub 2021 Dec 25. PMID 34963087
- [Background] Bayala B, Bassole IH, Gnoula C, Nebie R, Yonli A, Morel L, Figueredo G, Nikiema JB, Lobaccaro JM, Simpore J. Chemical composition, antioxidant, anti-inflammatory and anti-proliferative activities of essential oils of plants from Burkina Faso. PLoS One. 2014 Mar 24;9(3):e92122. doi: 10.1371/journal.pone.0092122. eCollection 2014. PMID 24662935
- [Background] Peterfalvi A, Miko E, Nagy T, Reger B, Simon D, Miseta A, Czeh B, Szereday L. Much More Than a Pleasant Scent: A Review on Essential Oils Supporting the Immune System. Molecules. 2019 Dec 11;24(24):4530. doi: 10.3390/molecules24244530. PMID 31835699
- [Background] Zhao ZJ, Sun YL, Ruan XF. Bornyl acetate: A promising agent in phytomedicine for inflammation and immune modulation. Phytomedicine. 2023 Jun;114:154781. doi: 10.1016/j.phymed.2023.154781. Epub 2023 Mar 22. PMID 37028250
- [Background] Zhang Z, Liu Q, Wen P, Zhang J, Rao X, Zhou Z, Zhang H, He X, Li J, Zhou Z, Xu X, Zhang X, Luo R, Lv G, Li H, Cao P, Wang L, Xu F. Activation of the dopaminergic pathway from VTA to the medial olfactory tubercle generates odor-preference and reward. Elife. 2017 Dec 18;6:e25423. doi: 10.7554/eLife.25423. PMID 29251597
- [Background] Bhimani RV, Yates R, Bass CE, Park J. Distinct limbic dopamine regulation across olfactory-tubercle subregions through integration of in vivo fast-scan cyclic voltammetry and optogenetics. J Neurochem. 2022 Apr;161(1):53-68. doi: 10.1111/jnc.15577. Epub 2022 Feb 5. PMID 35061915
- [Background] Ben-Shaanan TL, Schiller M, Azulay-Debby H, Korin B, Boshnak N, Koren T, Krot M, Shakya J, Rahat MA, Hakim F, Rolls A. Modulation of anti-tumor immunity by the brain's reward system. Nat Commun. 2018 Jul 13;9(1):2723. doi: 10.1038/s41467-018-05283-5. PMID 30006573
- [Background] Kite SM, Maher EJ, Anderson K, Young T, Young J, Wood J, Howells N, Bradburn J. Development of an aromatherapy service at a Cancer Centre. Palliat Med. 1998 May;12(3):171-80. doi: 10.1191/026921698671135743. PMID 9743836
- [Background] Deng C, Xie Y, Liu Y, Li Y, Xiao Y. Aromatherapy Plus Music Therapy Improve Pain Intensity and Anxiety Scores in Patients With Breast Cancer During Perioperative Periods: A Randomized Controlled Trial. Clin Breast Cancer. 2022 Feb;22(2):115-120. doi: 10.1016/j.clbc.2021.05.006. Epub 2021 May 20. PMID 34134947